CLINICAL TRIAL: NCT04429087
Title: A First-In-human Phase I, Non-randomized, Open-label, Multi-center Dose Escalation Trial of BI 764532 Administered by Parenteral Route in Patients With Small Cell Lung Carcinoma and Other Neuroendocrine Neoplasms Expressing DLL3
Brief Title: A Study to Test Different Doses of BI 764532 in Patients With Small Cell Lung Cancer and Other Neuroendocrine Tumours That Are Positive for DLL3
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1438-0001; 2019-000729-31 (EudraCT Number)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Patients With Small Cell Lung Carcinoma and Other Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: BI 764532 (Experimental)
  Interventions: Drug: BI 764532 - parenteral 1
- Arm 2: BI 764532 (Experimental)
  Interventions: Drug: BI 764532 - parenteral 2

INTERVENTIONS:
Drug: BI 764532 - parenteral 1 — BI 764532 - parenteral 1
  Other Names: Obrixtamig
  Arms: Arm 1: BI 764532
Drug: BI 764532 - parenteral 2 — BI 764532 - parenteral 2
  Other Names: Obrixtamig
  Arms: Arm 2: BI 764532

SUMMARY:
This study is open to adults with small cell lung cancer and other neuroendocrine cancers that are positive for the tumour marker delta-like 3 (DLL3). The study is in people with advanced cancer for whom previous treatment was not successful or no standard treatment exists.

The purpose of this study is to find out the highest dose of BI 764532 and the best treatment schedule that people can tolerate. BI 764532 is an antibody-like molecule (DLL3/CD3 bispecific) that may help the immune system fight cancer. In this study, BI 764532 is given to people for the first time. That means no clinical data are available for BI 764532.

Participants get BI 764532 either weekly or once every 3 weeks. If there is benefit for the participants and if they can tolerate it, the treatment is given for a maximum of 3 years. During this time, participants visit the study site about 20 times depending on the response to the treatment. Doctors record any unwanted effects and regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated, written informed consent form (ICF2, ICF3 or ICF4) in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) - Good Clinical Practice (GCP) and local legislation prior to any trial-specific procedures, sampling, or analyses.
* Locally advanced or metastatic cancer not amenable to curative treatment; of following histologies:

  * Small cell lung carcinoma (SCLC)
  * Large cells neuroendocrine lung carcinoma (LCNEC)
  * Neuroendocrine carcinoma (NEC) or small cell carcinoma of any other origin
  * Tumours must be positive for DLL3 expression (on archived tissue or instudy fresh biopsy) according to central pathology review in order to start BI 764532
  * Patients with tumours with mixed histologies for any above type are eligible only if neuroendocrine carcinoma/small tumor cells component is predominant and represent at least 50% of the overall tumour tissue.
* For back-fill cohorts only: patient has agreed to and signed an IC to provide mandatory pre-treatment and on-treatment fresh tumor biopsy.
* Patient has failed or is not eligible for available standard therapies according to local guidelines. Standard therapies should include at least one line of chemotherapy that should include platinum for patients with small cells carcinoma tumors histologies.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* At least one evaluable lesion outside of CNS as defined per modified Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Subjects with brain metastases are eligible provided they meet the following criteria:

  * Radiotherapy or surgery for brain metastases was completed at least 2 weeks prior to the first administration of BI 764532
  * Patient is off steroids for at least 7 days (physiologic doses of steroids are permitted), and the patient is off anti-epileptic drugs for at least 7 days or on stable doses of anti-epileptic drugs for malignant Central Nervous System (CNS) disease.
* Adequate liver, bone marrow and renal organ function Further inclusion criteria apply.

Exclusion Criteria:

* Previous treatment with T cell Engager (TcE) or cell therapies targeting DLL3. Other DLL3 targeting agents (like Rovalpituzumab tesirine (RovaT)) are allowed only if DLL3 positivity is documented after completion of treatment with DLL3 targeting agent in post-treatment biopsy.
* Anticoagulant treatment that cannot be safely interrupted based on opinion of the investigator if medically needed (e.g. biopsy).
* Persistent toxicity from previous treatments that has not resolved to = Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 (except for alopecia, CTCAE Grade 2 neuropathy, asthenia/fatigue or grade 2 endocrinopathies controlled by replacement therapy).
* Patient has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of BI 764532. Physiological replacement of steroids is allowed.
* Prior anti-cancer therapy:

  * Patients who have been treated with any other anti-cancer drug within 3 weeks or within 5 half-life periods (whichever is shorter) prior to first administration of BI 764532.
  * Patients who have been treated with extensive field radiotherapy including whole brain irradiation within 2 weeks prior to first administration of BI 764532.
* Other active malignancy that could interfere with the prognosis and treatment of the disease of the study.
* Major surgery within 28 days of first dose BI 764532.
* Women who are pregnant (including those who are considered to be possibly pregnant based on the investigator's clinical judgement), nursing/breast feeding or who plan to become pregnant or nurse while in the trial or within 35 days after the last dose of study treatment.
* Active infection that requires medical therapy or other clinically significant intervention or within 2 weeks prior to study entry confirmed (PCR test or other applicable test as per local requirements) or suspected SARS-CoV-2 infection or close contact with an individual with confirmed SARS-CoV-2 infection.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Arm 1 and Arm 2: Maximum tolerated dose (MTD) | up to 36 months
  Maximum tolerated dose (MTD) in any studied regimen defined as the highest dose with less than 25% risk of the true Dose Limiting Toxicity (DLT) rate being equal or above 33% during the MTD evaluation period. Separate MTDs will be determined for each Regimen.
Arm 1 and Arm 2: Number of patients with DLTs in the MTD evaluation period | up to 36 months

SECONDARY OUTCOMES:
Arm 1 and Arm 2: Maximum measured concentration (Cmax) of BI 764532 | up to 36 months
Arm 1 and Arm 2: Area under the concentration-time curve (AUCτ) of the analyte over a uniform dosing interval τ | up to 36 months
Arm 1 and Arm 2: Objective response based on RECIST 1.1 criteria in patients with measurable disease | up to 36 months
  Objective response based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in patients with measurable disease

CONTACTS AND LOCATIONS:
Locations (12):
- United States (4):
  - Winship Cancer Institute, Atlanta, Georgia
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Germany (3):
  - Universitätsklinikum Köln (AöR), Cologne
  - Technische Universität Dresden, Dresden
  - Universitätsklinikum Würzburg AÖR, Würzburg
- National Cancer Center Hospital East, Chiba, Kashiwa, Japan
- Spain (4):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario De Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Wermke M, Felip E, Gambardella V, Kuboki Y, Morgensztern D, Hamed ZO, Liu M, Studeny M, Owonikoko TK. Phase I trial of the DLL3/CD3 bispecific T-cell engager BI 764532 in DLL3-positive small-cell lung cancer and neuroendocrine carcinomas. Future Oncol. 2022 Aug;18(24):2639-2649. doi: 10.2217/fon-2022-0196. Epub 2022 Jul 11. PMID 35815644
- See also: Related Info — https://www.mystudywindow.com